CLINICAL TRIAL: NCT04518202
Title: Transdermal Lidocaine for Pain Control During Diagnostic Office Hysteroscopy: a Randomized Controlled Trial
Brief Title: Transdermal Lidocaine for Pain Control During Diagnostic Office Hysteroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/296/3/19
Record Dates: First submitted 2020-08-15; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Intervention Model Description: double blinded randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blinded randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine patch (Experimental): 5% lidocaine patch applied at 6 hours before the scheduled office hysteroscopy.
  Interventions: Drug: lidocaine patch
- Sham patch (Placebo Comparator): Sham patch applied at 6 hours before the scheduled office hysteroscopy.
  Interventions: Drug: Sham patch

INTERVENTIONS:
Drug: lidocaine patch — 5% lidocaine patch applied at 6 hours before the scheduled office hysteroscopy.
  Other Names: Experimental
  Arms: lidocaine patch
Drug: Sham patch — Sham patch containing no study medication applied at 6 hours before the scheduled office hysteroscopy.
  Other Names: Placebo Comparator
  Arms: Sham patch

SUMMARY:
To compare the effectiveness of Transdermal Lidocaine for Pain Control During Diagnostic Office Hysteroscopy

DETAILED DESCRIPTION:
hysteroscopy is commonly used in the diagnosis and treatment of intrauterine lesions such as polyps, ﬁbroids, septa, and adhesions, and in the presence of abnormal bleeding and during the removal of an intrauterine device or foreign body. Cervical ripening is made possible by the use of medication through different routes.

ELIGIBILITY:
Inclusion Criteria:

* patients with an indication for ofﬁce hysteroscopy

Exclusion Criteria:

* patient refuse to participant
* contraindication for lidocaine patch

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — patients with an indication for ofﬁce hysteroscopy
Enrollment: 200 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity will be assessed by visual analogue scale | 10 minutes
  Pain intensity will be assessed by visual analogue scale 30 minutes after the procedure. Visual analogue scale ranging from 0 to 10

SECONDARY OUTCOMES:
Operative time | 15 minutes
  From the introduction of hysteroscope into the vagina till compilation of hysteroscopic examination

CONTACTS AND LOCATIONS:
Overall Officials: nahla w Shady, md, Study Chair — Aswan universirty
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No